CLINICAL TRIAL: NCT04973475
Title: Prospective Clinical Trials on Clinical Outcomes of Indocyanine Green Tracer Using in Laparoscopic Distal Gastrectomy With Lymph Node Dissection for Early Gastric Cancer
Brief Title: Indocyanine Green Tracer Using in Laparoscopic Distal Gastrectomy for Early Gastric Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Professor, Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUGES-023
Record Dates: First submitted 2021-07-13; First posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Early Gastric Cancer; Indocyanine Green; Lymph Node Dissection
Keywords: Stomach Neoplasms; Indocyanine Green Tracer; Laparoscopic Distal Gastrectomy; Lymph Node Dissection
MeSH Terms: conditions — Stomach Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Indocyanine Green Tracer (Experimental): Indocyanine Green Tracer will be used in laparoscopic distal gastrectomy with lymph node dissection for gastric adenocarcinoma.
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — Laparoscopic distal gastrectomy with lymph node dissection for early gastric cancer using Indocyanine Green Tracer
  Other Names: ICG

SUMMARY:
This study aims to explore the value of indocyanine green (ICG) in laparoscopic distal gastrectomy with lymph node dissection for early gastric cancer.The patients with early gastric adenocarcinoma (cT1, N-/+, M0) will be studied.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will receiving injection of indocyanine greenat 8 points around the primary tumor with gastroscope 1 day before surgery. During the operation, laparoscopic gastrectomy and perigastric lymph node dissection were performed under ICG imaging equipment. After the surgical specimens were isolated, under the fluorescent illumination of the ICG imaging equipment, the lymph nodes that showed fluorescence and the lymph nodes that did not show fluorescence were collected from each LN station.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 75 years
2. Primary gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by endoscopic biopsy
3. Clinical stage tumor T1 (cT1), N0/+, M0 at preoperative evaluation according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual Eighth Edition. Preoperative staging was made by conducting mandatory computed tomography (CT) scans and an optional endoscopic ultrasound
4. No distant metastasis, no direct invasion of pancreas, spleen or other organs nearby in the preoperative examinations
5. Tumor located in the lower third of the stomach, expected to receive radical distal gastrectomy
6. Performance status of 0 or 1 on Eastern Cooperative Oncology Group scale (ECOG)
7. American Society of Anesthesiology score (ASA) class I, II, or III
8. Written informed consent

Exclusion Criteria:

1. Women during pregnancy or breast-feeding
2. Severe mental disorder
3. History of previous upper abdominal surgery (except laparoscopic cholecystectomy)
4. History of previous gastrectomy, endoscopic mucosal resection or endoscopic submucosal dissection
5. Enlarged or bulky regional lymph node diameter over 3cm by preoperative imaging
6. History of other malignant disease within past five years
7. History of previous neoadjuvant chemotherapy or radiotherapy
8. History of unstable angina or myocardial infarction within past six months
9. History of cerebrovascular accident within past six months
10. History of continuous systematic administration of corticosteroids within one month
11. Requirement of simultaneous surgery for other disease
12. Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer
13. Forced expiratory volume in 1 second (FEV1)<50% of predicted values
14. Rejection of laparoscopic resection
15. Preoperatively confirmed tumors invading the dentate line or duodenum
16. History of allergy to iodine agents
17. Tumor located in the upper third of the stomach, expected to receive radical total gastrectomy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
False negative rate | One month after surgery
  The number of positive lymph nodes in not fluorescent lymph nodes is divided by the number of total not fluorescent lymph nodes

SECONDARY OUTCOMES:
True positive rate | One month after surgery
  The number of positive lymph nodes in fluorescent lymph nodes is divided by the number of total fluorescent lymph nodes
False positive rate | One month after surgery
  The number of negative lymph nodes in fluorescent lymph nodes is divided by the number of total fluorescent lymph nodes
True negative rate | One month after surgery
  The number of negative lymph nodes in not fluorescent lymph nodes is divided by the number of total not fluorescent lymph nodes
Total number of retrieved lymph nodes | One month after surgery
  Total number of retrieved lymph nodes
Lymph node noncompliance rate | One month after surgery
  Lymph node noncompliance was defined as the absence of lymph nodes that should have been excised from more than 1 lymph node station. Major lymph node noncompliance was defined as more than 2 intended lymph node stations that were not removed.
Number of Metastasis Lymph Nodes | One month after surgery
  Number of Metastasis Lymph Nodes
Metastasis rate of lymph node | One month after surgery
  Metastasis rate of lymph node
Morbidity and mortality rates | One month after surgery
  This is for the early postoperative complication and mortality, which defined as the event observed within 30 days after surgery.
3-year overall survival rate | 36 months
  3-year overall survival rate
3-year disease free survival rate | 36 months
  3-year disease free survival rate
3-year recurrence pattern | 36 months
  Recurrence patterns are classified into five categories at the time of first diagnosis: locoregional, hematogenous, peritoneal, distant lymph node, and mixed type.
Intraoperative morbidity rates | 1 day
  The intraoperative postoperative morbidity rates are defined as the rates of event observed within operation.
Time to first ambulation | 30 days
  Time to first ambulation in hours is used to assess the postoperative recovery course.
Time to first flatus | 30 days
  Time to first flatus in days is used to assess the postoperative recovery course.
Time to first liquid diet | 30 days
  Time to first liquid diet in days is used to assess the postoperative recovery course.
Time to first soft diet | 30 days
  Time to first soft diet in days is used to assess the postoperative recovery course.
Duration of postoperative hospital stay | 30 days
  Duration of postoperative hospital stay in days is used to assess the postoperative recovery course.
The variation of white blood cell count | Preoperative 3 days and postoperative 1, 3, and 5 days
  The values of white blood cell count from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.
The variation of hemoglobin | Preoperative 3 days and postoperative 1, 3, and 5 days
  The values of hemoglobin in gram/liter from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.
The variation of C-reactive protein | Preoperative 3 days and postoperative 1, 3, and 5 days
  The variation of C-reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Ming Huang, MD, Study Chair — Fujian Medical University Union Hospital
Locations (1):
- Department of Gastric Surgery, Fuzhou, Fujian, China

REFERENCES:
- [Background] Fock KM. Review article: the epidemiology and prevention of gastric cancer. Aliment Pharmacol Ther. 2014 Aug;40(3):250-60. doi: 10.1111/apt.12814. Epub 2014 Jun 10. PMID 24912650
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Msika S, Chastang C, Houry S, Lacaine F, Huguier M. Lymph node involvement as the only prognostic factor in curative resected gastric carcinoma: a multivariate analysis. World J Surg. 1989 Jan-Feb;13(1):118-23; discussion 123. doi: 10.1007/BF01671171. PMID 2471364
- [Background] Maruyama K, Gunven P, Okabayashi K, Sasako M, Kinoshita T. Lymph node metastases of gastric cancer. General pattern in 1931 patients. Ann Surg. 1989 Nov;210(5):596-602. doi: 10.1097/00000658-198911000-00005. PMID 2818028
- [Background] Zhang YX, Yang K. Significance of nodal dissection and nodal positivity in gastric cancer. Transl Gastroenterol Hepatol. 2020 Apr 5;5:17. doi: 10.21037/tgh.2019.09.13. eCollection 2020. PMID 32258521
- [Background] Mocellin S. The Effect of Lymph Node Dissection on the Survival of Patients With Operable Gastric Carcinoma. JAMA Oncol. 2016 Oct 1;2(10):1363-1364. doi: 10.1001/jamaoncol.2016.2044. PMID 27442439
- [Background] Japanese Gastric Cancer Association. Japanese gastric cancer treatment guidelines 2018 (5th edition). Gastric Cancer. 2021 Jan;24(1):1-21. doi: 10.1007/s10120-020-01042-y. Epub 2020 Feb 14. No abstract available. PMID 32060757
- [Background] Sasako M, McCulloch P, Kinoshita T, Maruyama K. New method to evaluate the therapeutic value of lymph node dissection for gastric cancer. Br J Surg. 1995 Mar;82(3):346-51. doi: 10.1002/bjs.1800820321. PMID 7796005
- [Background] Kurokawa Y, Takeuchi H, Doki Y, Mine S, Terashima M, Yasuda T, Yoshida K, Daiko H, Sakuramoto S, Yoshikawa T, Kunisaki C, Seto Y, Tamura S, Shimokawa T, Sano T, Kitagawa Y. Mapping of Lymph Node Metastasis From Esophagogastric Junction Tumors: A Prospective Nationwide Multicenter Study. Ann Surg. 2021 Jul 1;274(1):120-127. doi: 10.1097/SLA.0000000000003499. PMID 31404008
- [Background] Baiocchi GL, Giacopuzzi S, Reim D, Piessen G, Costa PMD, Reynolds JV, Meyer HJ, Morgagni P, Gockel I, Santos LL, Jensen LS, Murphy T, D'Ugo D, Rosati R, Fumagalli Romario U, Degiuli M, Kielan W, Monig S, Kolodziejczyk P, Polkowski W, Pera M, Schneider PM, Wijnhoven B, de Steur WO, Gisbertz SS, Hartgrink H, van Sandick JW, Botticini M, Holscher AH, Allum W, De Manzoni G. Incidence and Grading of Complications After Gastrectomy for Cancer Using the GASTRODATA Registry: A European Retrospective Observational Study. Ann Surg. 2020 Nov;272(5):807-813. doi: 10.1097/SLA.0000000000004341. PMID 32925254
- [Background] Han SU, Hur H, Lee HJ, Cho GS, Kim MC, Park YK, Kim W, Hyung WJ; Korean Laparoendoscopic Gastrointestinal Surgery Study (KLASS) Group. Surgeon Quality Control and Standardization of D2 Lymphadenectomy for Gastric Cancer: A Prospective Multicenter Observational Study (KLASS-02-QC). Ann Surg. 2021 Feb 1;273(2):315-324. doi: 10.1097/SLA.0000000000003883. PMID 33064386
- [Background] Liu M, Xing J, Xu K, Yuan P, Cui M, Zhang C, Yang H, Yao Z, Zhang N, Tan F, Su X. Application of Near-Infrared Fluorescence Imaging with Indocyanine Green in Totally Laparoscopic Distal Gastrectomy. J Gastric Cancer. 2020 Sep;20(3):290-299. doi: 10.5230/jgc.2020.20.e25. Epub 2020 Aug 31. PMID 33024585
- [Background] Roh CK, Choi S, Seo WJ, Cho M, Son T, Kim HI, Hyung WJ. Indocyanine green fluorescence lymphography during gastrectomy after initial endoscopic submucosal dissection for early gastric cancer. Br J Surg. 2020 May;107(6):712-719. doi: 10.1002/bjs.11438. Epub 2020 Feb 7. PMID 32031248
- [Background] Cianchi F, Indennitate G, Paoli B, Ortolani M, Lami G, Manetti N, Tarantino O, Messeri S, Foppa C, Badii B, Novelli L, Skalamera I, Nelli T, Coratti F, Perigli G, Staderini F. The Clinical Value of Fluorescent Lymphography with Indocyanine Green During Robotic Surgery for Gastric Cancer: a Matched Cohort Study. J Gastrointest Surg. 2020 Oct;24(10):2197-2203. doi: 10.1007/s11605-019-04382-y. Epub 2019 Sep 4. PMID 31485904